CLINICAL TRIAL: NCT01322529
Title: Preterm Birth in Nulliparous Women: An Understudied Population at Great Risk
Brief Title: Nulliparous Pregnancy Outcomes Study: Monitoring Mothers-to-be
Acronym: nuMoM2b
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Office of Research on Women's Health (ORWH) (NIH)
Responsible Party: Sponsor
Other Study IDs: NICHD-nuMoM2b-001; 1U10HD063036-01 (NIH); 1U10HD063072-01 (NIH); 1U10HD063047-01 (NIH); 1U10HD063037-01 (NIH); 1U10HD063041-01 (NIH); 1U10HD063020-01 (NIH); 1U10HD063046-01 (NIH); 1U10HD063048-01 (NIH); 1U10HD063053-01 (NIH)
Record Dates: First submitted 2011-03-10; First posted 2011-03-24 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Pregnancy; Pregnancy Complications
Keywords: nulliparity; pregnant women; pregnancy outcomes; pregnancy complications
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum, blood plasma, maternal deoxyribonucleic acid (DNA), urine supernatant, urine cell pellet, cervico-vaginal fluid, bacterial vaginosis (BV) slide, cord blood (fetal DNA), cord blood serum, placenta, fetal membranes, umbilical cord segment, placenta and umbilical cord, chorionic villi and maternal decidua from clinical chorionic villus sampling (CVS), amniotic fluid supernatant and cell pellet from clinical amniocentesis.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Forty percent of pregnant women in the United States are women who have never given birth. As a group, they sometimes have complications with their pregnancy, but there is no information from a previous pregnancy to identify who might have a problem. Very little research has been done with this group. The Nulliparous Pregnancy Outcomes Study: Monitoring Mothers-to-be (nuMoM2b) is collecting data from a diverse population of about 10,000 women who are having their first baby and are carrying only one baby. The women are enrolled early in pregnancy and undergo research assessments four times during their pregnancies. Data are collected through interviews, self-completed data forms, clinical measurements, ultrasound, and collection and storage of blood samples, urine samples, and fluid from the vagina and cervix. Some information comes from medical records. A subset of women may be asked to participate in substudies collecting information on sleep breathing, sleep patterns and quality, or other areas possibly related to birth outcomes. The goal of the research is to find ways to identify women in this group who might develop a problem with their pregnancy and use this information to improve the health of pregnant women and their babies in the future. The study is focusing on pregnancy problems like high blood pressure, babies that are born much too early and very small babies.

DETAILED DESCRIPTION:
The Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) established the Nulliparous Pregnancy Outcomes Study: Monitoring Mothers-to-be (nuMoM2b) to study women for whom the current pregnancy will lead to their first delivery (nulliparas). About 40% of pregnant women in the United States are nulliparas. Because little or no information from previous pregnancy outcomes is available to guide assignment of risk or mitigating interventions, adverse pregnancy outcomes in nulliparas are especially unpredictable. The underlying mechanisms of adverse pregnancy outcomes such as preterm birth, preeclampsia, fetal growth restriction and stillbirth are interrelated and therefore will be evaluated as part of this study. The information gained will benefit women who are pregnant or who are considering pregnancy and their physicians. In addition, the knowledge will support future research aimed at improving care and health outcomes for a critical group of at-risk women who are currently understudied.

The study is a prospective cohort study of a racially/ethnically/geographically diverse population of 10,038 nulliparous women with singleton gestations. The women undergo intensive research assessments during the course of their pregnancies to study the mechanisms for and prediction of adverse pregnancy outcomes (APOs) in women in their first pregnancy. The APOs of primary interest are preterm birth, preeclampsia and fetal growth restriction.

The goals of the study are to 1) determine maternal characteristics, including genetics, epigenetics, and physiological response to pregnancy as well as environmental factors that influence and/or predict adverse pregnancy outcome; 2) identify specific aspects of placental development and function that lead to adverse pregnancy outcome; and 3) characterize genetic, growth, and developmental parameters of the fetus that are associated with adverse pregnancy outcome.

Eight academic medical centers or sites had primary responsibility for enrollment and follow-up of study participants. Several of these sites collected data through additional academic research centers or nearby hospitals (subsites). A Data Coordinating and Analysis Center (DCAC) provided input to the protocol, manages the data, and analyzes the data. Investigators from these institutions have established a partnership with NICHD staff to develop and implement the study protocol and ancillary studies that acquire and analyze data to identify biomarkers and understand the mechanism and prediction of preterm birth and other adverse pregnancy outcomes.

Nulliparous women with an in utero singleton gestation between 6 weeks 0 days and 13 weeks 6 days of pregnancy were recruited through the eight clinical sites and their subsites. Mechanisms were created in the various prenatal clinics associated with the sites to identify eligible nulliparous women with singleton pregnancies. Once enrolled, a participant was followed for the duration of her pregnancy by research staff at the clinical site. Study visits were scheduled at four times during the pregnancy: 6 weeks 0 days through 13 weeks 6 days estimated gestational age (EGA), 16 weeks 0 days through 21 weeks 6 days EGA, 22 weeks 0 days through 29 weeks 6 days EGA, and at the time of delivery. Data were collected through personal interview, self-administered questionnaires, clinical measurement, chart abstraction, and collection of biological specimens (blood, urine, cervico-vaginal fluid). Additional data (i.e., sleep breathing assessments, actigraphy, fetal adrenal gland measurements) were collected through ancillary research studies on subsets of the enrolled women. The set-ups for screening, enrollment and follow-up of participants varied by clinical site and subsite. However, in each setting, the clinical site staffs included study investigators, research nurses, research assistants and sonographers. Clinical site staffs were trained to interview participants, collect and process samples, conduct various research tests, and input data. Data are managed at the DCAC. Specimens are stored at the NICHD specimen repository for later analysis.

ELIGIBILITY:
Inclusion Criteria:

* Nullipara - Pregnant women with no prior pregnancy lasting 20 weeks 0 days or greater.
* Viable singleton gestation - a single living fetus with fetal cardiac activity at the most recent ultrasound before enrollment
* Between 6 weeks 0 days and 13 weeks 6 days project estimated gestational age (EGA) at first study visit.
* Intend to deliver at a participating hospital.

Exclusion Criteria:

* Participant age <13 years.
* History of 3 or more spontaneous abortions.
* Fetal malformation evident at or before enrollment that is likely lethal (e.g., anencephaly, hydrops, diffuse subcutaneous edema or cystic hygroma, ectopic cordis, encephalocele).
* Known fetal aneuploidy (based on chorionic villus sampling).
* Surrogate pregnancy (donor oocyte pregnancy).
* Multifetal reduction.
* Participating in an intervention study that is anticipated to influence maternal or fetal morbidities/mortality unless it is determined before enrollment that the study code will be made available.
* Woman previously enrolled in this study, including those consented but delivered before 20 weeks 0 days gestation.
* Planned pregnancy termination.
* Unable to provide informed consent.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of a racially/ethnically/geographically diverse population of 10,038 nulliparous pregnant women with singleton gestations recruited through 8 participating clinical sites and their subsites.
Sampling Method: Non-Probability Sample
Enrollment: 10038 (Actual)
Dates: Start 2010-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Adverse pregnancy outcome | 42 weeks project estimated gestational age or less
  Delivery of a live born or stillborn infant due to any cause before 37 weeks 0 days project estimated gestational age, after the subject has been enrolled in the study.

SECONDARY OUTCOMES:
Preterm birth | 42 weeks project estimated gestational age or less
  Delivery of a liveborn or stillborn infant for any cause between 20 weeks 0 days and 36 weeks 6 days project estimated gestational age.
Spontaneous preterm birth | 42 weeks project estimated gestational age or less
  Delivery occurring subsequent to spontaneous onset of preterm labor OR preterm Premature Rupture of the Membranes (preterm PROM) OR fetal membrane prolapse, regardless of subsequent labor augmentation or cesarean delivery.
Indicated preterm birth | 42 weeks project estimated gestational age or less
  Delivery following induction or cesarean delivery at less than 37 weeks 0 days gestation for one or more conditions that the woman's caregiver determines to threaten the health/life of the mother or fetus. The primary diagnoses associated with indicated preterm birth are categorized as follows: pregnancy associated hypertension, fetal growth restriction, abruptio placentae, placenta previa, chorioamnionitis, abnormal fetal testing, congenital fetal anomaly(ies), maternal medical condition, other, not documented.
Spontaneous pregnancy loss less than 20 weeks | 42 weeks project estimated gestational age or less
  Fetal death leading to vaginal delivery or dilatation and curettage/evacuation, or spontaneous expulsion of a liveborn fetus due to any cause before 20 weeks 0 days project EGA.

CONTACTS AND LOCATIONS:
Overall Officials: George Saade, M.D., Study Chair — University of Texas; Brian M Mercer, M.D., Principal Investigator — Case Western Reserve University; Ronald Wapner, M.D., Principal Investigator — Columbia University; David M Haas, M.D., M.S., Principal Investigator — Indiana University; Hyagriv N Simhan, MD, MSCR, Principal Investigator — Magee-Women's Hospital - University of Pittsburgh; William Grobman, M.D., M.B.A., Principal Investigator — Northwestern University; Deborah A Wing, M.D., Principal Investigator — University of California, Irvine; Samuel Parry, M.D., Principal Investigator — University of Pennsylvania; Robert M Silver, M.D., Principal Investigator — University of Utah; Cora (Corette) B Parker, MSPH, DrPH, Principal Investigator — RTI International
Locations (17):
- United States (17):
  - Fountain Valley Regional Hospital and Medical Center- UCI MFM private practice, Fountain Valley, California
  - Long Beach Memorial Medical Center, Women's and Children's Hospital - Women's Perinatal Group, OB Clinic, Long Beach, California
  - University of California, Irvine, Medical Center - Prenatal care clinics and private practice, Orange, California
  - Christiana Care Health Systems, Newark, Delaware
  - Northwestern University, Chicago, Illinois
  - Indiana University School of Medicine OB/GYN, Indianapolis, Indiana
  - Columbia University Medical Center- Department of Obstetrics and Gynecology Division of Maternal Fetal Medicine, New York, New York
  - Case Western Reserve University, MetroHealth Medical Center, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - West Penn Allegheny Health System, Pittsburgh, Pennsylvania
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - McKay Dee Hospital, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - University of Utah, Salt Lake City, Utah
  - Intermountain Medical Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided
Date will be made available to authorized researchers in the future through a yet to be determined government repository.

REFERENCES:
- [Background] Haas DM, Parker CB, Wing DA, Parry S, Grobman WA, Mercer BM, Simhan HN, Hoffman MK, Silver RM, Wadhwa P, Iams JD, Koch MA, Caritis SN, Wapner RJ, Esplin MS, Elovitz MA, Foroud T, Peaceman AM, Saade GR, Willinger M, Reddy UM; NuMoM2b study. A description of the methods of the Nulliparous Pregnancy Outcomes Study: monitoring mothers-to-be (nuMoM2b). Am J Obstet Gynecol. 2015 Apr;212(4):539.e1-539.e24. doi: 10.1016/j.ajog.2015.01.019. Epub 2015 Jan 31. PMID 25648779
- [Background] Facco FL, Parker CB, Reddy UM, Silver RM, Louis JM, Basner RC, Chung JH, Schubert FP, Pien GW, Redline S, Mobley DR, Koch MA, Simhan HN, Nhan-Chang CL, Parry S, Grobman WA, Haas DM, Wing DA, Mercer BM, Saade GR, Zee PC. NuMoM2b Sleep-Disordered Breathing study: objectives and methods. Am J Obstet Gynecol. 2015 Apr;212(4):542.e1-127. doi: 10.1016/j.ajog.2015.01.021. Epub 2015 Mar 4. PMID 25746730
- [Derived] Haas DM, Moss K, Faysal H, Yee LM, Silver RM, Grobman WA. First trimester urine glyphosate concentrations and gestational diabetes in nulliparas: a nested case-control study. Environ Health. 2025 Oct 7;24(1):71. doi: 10.1186/s12940-025-01183-6. PMID 41057879
- [Derived] Venkatesh KK, Yee LM, Johnson J, Wu J, McNeil B, Mercer B, Simhan H, Reddy UM, Silver RM, Parry S, Saade G, Chung J, Wapner R, Lynch CD, Grobman WA. Neighborhood Socioeconomic Disadvantage and Abnormal Birth Weight. Obstet Gynecol. 2023 Nov 1;142(5):1199-1207. doi: 10.1097/AOG.0000000000005384. Epub 2023 Sep 28. PMID 37769319
- [Derived] Haas DM, Yang Z, Parker CB, Chung J, Parry S, Grobman WA, Mercer BM, Simhan HN, Silver RM, Wapner RJ, Saade GR, Greenland P, Merz NB, Reddy UM, Pemberton VL; nuMoM2b study and the nuMoM2b Heart Health Study. Factors associated with duration of breastfeeding in women giving birth for the first time. BMC Pregnancy Childbirth. 2022 Sep 22;22(1):722. doi: 10.1186/s12884-022-05038-7. PMID 36138368
- [Derived] Beck C, Allshouse A, Silver RM, Grobman WA, Simhan H, Haas D, Reddy UM, Blue NR. High early pregnancy body mass index is associated with alterations in first- and second-trimester angiogenic biomarkers. Am J Obstet Gynecol MFM. 2022 May;4(3):100614. doi: 10.1016/j.ajogmf.2022.100614. Epub 2022 Mar 10. PMID 35283347
- [Derived] Blue NR, Allshouse AA, Grobman WA, Day RC, Haas DM, Simhan HN, Parry S, Saade GR, Silver RM. Developing a predictive model for perinatal morbidity among small for gestational age infants. J Matern Fetal Neonatal Med. 2022 Dec;35(25):8462-8471. doi: 10.1080/14767058.2021.1980533. Epub 2021 Sep 28. PMID 34582307
- [Derived] Miller ES, Saade GR, Simhan HN, Monk C, Haas DM, Silver RM, Mercer BM, Parry S, Wing DA, Reddy UM, Grobman WA. Trajectories of antenatal depression and adverse pregnancy outcomes. Am J Obstet Gynecol. 2022 Jan;226(1):108.e1-108.e9. doi: 10.1016/j.ajog.2021.07.007. Epub 2021 Jul 17. PMID 34280383
- [Derived] Dude AM, Plunkett B, Grobman W, Scifres CM, Mercer BM, Parry S, Silver RM, Wapner R, Wing DA, Saade G, Reddy U, Iams J, Simhan H, Kominiarek MA. The association between personal weight gain goals, provider recommendations, and appropriate gestational weight gain. Am J Obstet Gynecol MFM. 2020 Nov;2(4):100231. doi: 10.1016/j.ajogmf.2020.100231. Epub 2020 Sep 22. PMID 33345934
- [Derived] Haas DM, Mahnke B, Yang Z, Guise D, Daggy J, Simhan HN, Silver RM, Grobman WA, Wapner RJ, Makhoul J, Parry S, Mercer BM, Saade GR. Profile of Reported Alcohol, Tobacco, and Recreational Drug Use in Nulliparous Women. Obstet Gynecol. 2020 Jun;135(6):1281-1288. doi: 10.1097/AOG.0000000000003826. PMID 32459419
- [Derived] Premkumar A, Debbink MP, Silver RM, Haas DM, Simhan HN, Wing DA, Parry S, Mercer BM, Iams J, Reddy UM, Saade G, Grobman WA. Association of Acculturation With Adverse Pregnancy Outcomes. Obstet Gynecol. 2020 Feb;135(2):301-309. doi: 10.1097/AOG.0000000000003659. PMID 31923068
- [Derived] Haas DM, Marsh DJ, Dang DT, Parker CB, Wing DA, Simhan HN, Grobman WA, Mercer BM, Silver RM, Hoffman MK, Parry S, Iams JD, Caritis SN, Wapner RJ, Esplin MS, Elovitz MA, Peaceman AM, Chung J, Saade GR, Reddy UM. Prescription and Other Medication Use in Pregnancy. Obstet Gynecol. 2018 May;131(5):789-798. doi: 10.1097/AOG.0000000000002579. PMID 29630018
- [Derived] Michaliszyn SF, Sjaarda LA, Scifres C, Simhan H, Arslanian SA. Maternal excess gestational weight gain and infant waist circumference: a 2-y observational study. Pediatr Res. 2017 Jan;81(1-1):63-67. doi: 10.1038/pr.2016.174. Epub 2016 Sep 15. PMID 27632776